CLINICAL TRIAL: NCT06568757
Title: The Effect of Wet Cupping Therapy on Headache Severity and Disability in Patients Diagnosed With Migraine
Brief Title: The Effect of Wet Cupping Therapy on Headache and Migraine-related Disability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Sultan ÇEÇEN, Lecturer PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Wet Cupping Therapy
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Migraine-related Headache
Keywords: wet cupping; migraine; headache; disability
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wet Cupping Group (Experimental): The group that will receive wet cupping therapy-cupping application to the head and neck area in addition to medical treatment
  Interventions: Other: Wet Cupping
- Control Group (Active Comparator): The group that will not receive any treatment other than medical treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Wet Cupping — Wet cupping therapy will be applied once using disposable plastic vacuum cups to a total of 4 areas, which are recommended areas for headaches; cervical spine C7 (DU14 acupuncture point), bilateral T2-4 lateral spine (BL41-42 acupuncture point) and suboccipital region (FengFu DU-16 acupuncture point).
  Arms: Wet Cupping Group
Other: No intervention — No treatment will be applied to individuals and the routine medical treatment program will continue.
  Arms: Control Group

SUMMARY:
Objective: This study aims to investigate the effects of wet cupping therapy (cupping) applied once to the head and neck region on the severity of headache and disability in patients diagnosed with migraine.

Method: The research will be conducted as a pre-test-post-test, randomized controlled and qualitative study. Participants in the wet cupping group will receive wet cupping therapy using disposable plastic vacuum cups in a total of 4 regions including the cervical spine C7 (DU14 acupuncture point), bilateral T2-4 lateral spine (BL41-42 acupuncture point) and the suboccipital region (FengFu DU-16 acupuncture point). No intervention other than medical treatment will be applied to the control group. Patients in both groups will continue their routine treatments throughout the study. Before the intervention, the Patient Introduction Form, Wet Cupping Therapy Patient Feedback Form (pre-intervention) and Migraine Disability Assessment Scale (MIDAS) will be filled out. One month after the intervention, the Wet Cupping Therapy Patient Opinion Form (post-intervention) and the MIDAS will be re-evaluated after 3 months.

Results: Statistical analyses of the data will be performed using the Statistical Package for Social Sciences (Version 22.0, SPSS Inc., Chicago, IL, USA, License: Hitit University). Depending on the homogeneity of the data distribution, appropriate parametric or non-parametric tests will be applied for data evaluation.

DETAILED DESCRIPTION:
The cupping application, which has a very old history and varies in different countries and cultures, is preferred especially in Islamic geography as wet cupping application and in Far Eastern countries as dry cupping application. In dry cupping application, the cup material (plastic, glass, bamboo) is attached to the application area by creating negative pressure and the skin is swollen. Blood collection is not performed in this application. In wet cupping application, the application is started with dry cupping application and then superficial incisions are made on the skin in order to drain the blood from the skin and the cup is closed again. When some interstitial fluid is observed, the application is terminated. Although the mechanism of action of wet cupping application has not been fully explained, it is stated that it has neural, hematological, immunological, metabolic and psychological effects. In addition, all the effects of cupping are interrelated and neural effect is explained by the gate control theory.

Cupping application is added to the treatment of many diseases that affect different systems, especially hypertension, low back pain, hyperlipidemia. Migraine is one of these diseases.

Migraine, a chronic neurovascular disorder, is a disease characterized by moderate to severe headache attacks typically accompanied by nausea, vomiting, photophobia or phonophobia. Migraine, which ranks second among the diseases that cause disability worldwide, negatively affects the quality of life of individuals. In addition, migraine, which creates a great socioeconomic burden, is the most common disability-causing disorder in young women. Therefore, acute and prophylactic treatments for migraine are gaining importance in terms of improving the quality of life and reducing the burden. Although pharmacological treatment guidelines for migraine have been developed and updated, limitations arise due to excessive use, resistance and side effects in drug treatment. For this reason, many complementary and integrative treatment methods such as mindfulness meditation, yoga, tai chi, chiropractic, acupuncture, massage, phytotherapy, homeopathy, bloodletting and cupping are used in migraine treatment. There are a limited number of studies in the literature where cupping is applied in migraine treatment and its effect on pain intensity is evaluated. While all the study results found that cupping therapy reduces pain intensity, two studies found that it also reduces disability in addition to this result. According to the meta-analysis results of Seo et al. (2021), which included 6 randomized controlled trials (RCTs) from 218 studies, it was determined that cupping therapy reduces pain intensity and can significantly increase quality of life. However, it is stated that better designed RCTs are needed due to the low quality of evidence. Therefore, this study, which was planned to create evidence-based data for the literature, aims to examine the effect of cupping therapy on migraine-related disability and pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-65,
* Those who are literate, speak Turkish and have no communication problems,
* Those diagnosed with migraine according to the International Classification of Headache Disorders (ICHD-3),
* Those who have had headaches for the last three months and are receiving medical treatment for this reason,
* Those who want to have cupping therapy,
* Those who do not have any bleeding or coagulation disorders,
* Those who have not had wet cupping therapy in the last three months,
* Those who have a contraindication for wet cupping therapy (e.g. hemoglobin values below 9.5 gr/dl, INR below 1.5),
* Those who do not have a history of malignancy,
* Those who do not have an open wound in the application area,
* Those who do not have any psychiatric disorders

Exclusion Criteria:

* Patients with any incurable disease,
* Patients with a physical disability in the area where the application will be made,
* Patients with any skin disease in the area where the application will be made,
* Patients with large scar tissue in the area where the application will be made,
* Patients with a history of physical trauma in the area where the application will be made in the last three months,
* Patients with any peripheral vascular disease in the area where the application will be made,
* Patients who have used any complementary and integrative health application in the last three months,
* Patients who have received pain blockade treatment in the last year

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-23 (Estimated); Primary Completion 2024-10-24 (Estimated); Study Completion 2025-03-17 (Estimated)

PRIMARY OUTCOMES:
Wet Cupping Therapy Patient Opinion Form (Pre-Intervention) | Day 1
  It includes open-ended questions created by the researcher about how the patient's migraine headache affects his/her life and whether he/she believes in the effect of wet cupping in reducing pain.
Migraine Disability Assessment Scale (MIDAS) | Day 1
  It consists of 7 questions, the 1st, 3rd and 5th questions of which assess the days lost from school, work, housework or leisure activities due to headache in the last 3 months. The total MIDAS score is obtained by summing the first 5 questions. The total score is interpreted as 0-5 points as grade 1 (little or no restrictions), 6-10 points as grade 2 (mild or occasional restrictions), 11-20 points as grade 3 (moderate restrictions) and 21 or more points as grade 4 (severe restrictions).

SECONDARY OUTCOMES:
Wet Cupping Therapy Patient Opinion Form (Post-Intervention) | 1 months later
  It is a form created by the researcher and includes the questions, "Did wet cupping therapy reduce the intensity and frequency of pain?, What are the easy and difficult aspects of wet cupping therapy?, Were there any side effects of wet cupping therapy?"
Migraine Disability Assessment Scale (MIDAS) | 3 months later
  It consists of 7 questions, the 1st, 3rd and 5th questions of which assess the days lost from school, work, housework or leisure activities due to headache in the last 3 months. The total MIDAS score is obtained by summing the first 5 questions. The total score is interpreted as 0-5 points as grade 1 (little or no restrictions), 6-10 points as grade 2 (mild or occasional restrictions), 11-20 points as grade 3 (moderate restrictions) and 21 or more points as grade 4 (severe restrictions).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdulah DM, Mohammedsadiq HA, Mohammed AH. Effectiveness of wet cupping therapy on relieving pain in patients with chronic migraine: an observational study. J Complement Integr Med. 2021 Apr 1;18(3):569-577. doi: 10.1515/jcim-2020-0183. PMID 33793142